CLINICAL TRIAL: NCT05170828
Title: PRESERVE: A Multi-Center Trial Using Banked, Cryopreserved HLA-Mismatched Unrelated Donor Bone Marrow and Post-Transplantation Cyclophosphamide in Allogeneic Transplantation for Patients With Hematologic Malignancies
Brief Title: Cryopreserved MMUD BM With PTCy for Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in Study Design
Sponsor: Ossium Health, Inc. (Industry)
Collaborators: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRESERVE; NCT05068401 (obsolete NCT alias)
Record Dates: First submitted 2021-11-12; First posted 2021-12-28 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Acute Leukemia; Myelodysplastic Syndromes; T-lymphoblastic Lymphoma; Acute Lymphocytic Leukemia; Acute Myeloid Leukemia; Acute Biphenotypic Leukemia; Acute Undifferentiated Leukemia
Keywords: Leukemia; MDS; T-LBL; ALL; AML; ABL; AUL; Bone marrow transplant
MeSH Terms: conditions — Myelodysplastic Syndromes; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Busulfan; Mesna; Sirolimus; Mycophenolic Acid; Filgrastim; Granulocyte Colony-Stimulating Factor; Bone Marrow Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Regmin A (RIC) (Other): Pre-transplant conditioning treatment with Fludarabine, Cyclophosphamide, and Total Body Irradiation (TBI)
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total Body Irradiation; Drug: Mesna; Drug: Sirolimus; Drug: Mycophenolate Mofetil; Drug: Filgrastim; Procedure: Bone Marrow Transplant
- Regimen B (FIC) (Other): Pre-transplant conditioning treatment with Busulfan and Cyclophosphamide OR Fludarabine
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Busulfan; Drug: Mesna; Drug: Sirolimus; Drug: Mycophenolate Mofetil; Drug: Filgrastim; Procedure: Bone Marrow Transplant
- Regimen C (FIC) (Other): Pre-transplant conditioning treatment with Cyclophosphamide and Total Body Irradiation (TBI)
  Interventions: Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Drug: Mesna; Drug: Sirolimus; Drug: Mycophenolate Mofetil; Drug: Filgrastim; Procedure: Bone Marrow Transplant

INTERVENTIONS:
Drug: Cyclophosphamide — pre-transplant conditioning treatment
  Other Names: Cytoxan
Drug: Fludarabine — pre-transplant conditioning treatment
  Other Names: Fludara
  Arms: Regimen B (FIC); Regmin A (RIC)
Radiation: Total Body Irradiation — pre-transplant conditioning treatment
  Other Names: TBI
  Arms: Regimen C (FIC); Regmin A (RIC)
Drug: Busulfan — pre-transplant conditioning treatment
  Other Names: Busulfelx
  Arms: Regimen B (FIC)
Drug: Mesna — given with cyclophosphamide
  Other Names: Mesnex
Drug: Sirolimus — post-transplant treatment for GVHD
Drug: Mycophenolate Mofetil — post-transplant treatment for GVHD
  Other Names: MMF
Drug: Filgrastim — post-transplant treatment for GVHD
  Other Names: G-CSF
Drug: Cyclophosphamide — post-transplant treatment for GVHD
  Other Names: Cytoxan
Procedure: Bone Marrow Transplant — Transplant with investigational bone marrow product
  Other Names: Hematopoietic Stem Cell Transplant

SUMMARY:
Multicenter single arm study to assess the safety and efficacy of allogeneic transplantation using cryopreserved bone marrow from deceased MMUD and PTCy, sirolimus and MMF for GVHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged ≥ 18 and < 71 years (Note: HIV-negative subjects with MDS must be aged <50 at the time of signing the informed consent form)
* Diagnosed with
* Acute leukemias or T-lymphoblastic lymphoma (T-LBL) in 1st or subsequent CR
* Acute lymphocytic leukemia (ALL) or T-LBL as defined by the following:
* < 5% blasts in the bone marrow
* Normal maturation of all cellular components in the bone marrow
* No currently active extramedullary disease (EMD) (e.g., central nervous system (CNS), soft tissue disease)
* ANC ≥ 1,000/mm3
* Acute myeloid leukemia (AML) defined by the following:
* < 5% blasts in the bone marrow
* No blasts with Auer rods
* Normal maturation of all cellular components in the bone marrow
* No currently active EMD (e.g., CNS, soft tissue disease)
* ANC ≥ 1,000/mm3
* Acute biphenotypic leukemia (ABL)/Acute undifferentiated leukemia (AUL) defined by the following:
* < 5% blasts in the bone marrow
* Normal maturation of all cellular components in the bone marrow
* No currently active EMD (e.g., CNS, soft tissue disease)
* ANC ≥ 1,000/mm3
* Myleodysplastic Syndromes (MDS), fulfilling the following criteria:
* Subjects with de novo MDS who have or have previously had Intermediate-2 or High-risk disease as determined by the IPSS. Current Intermediate-2 or High- risk disease is not a requirement
* Subjects must have < 20% bone marrow blasts, assessed within 60 days of informed consent
* Subjects may have received prior therapy for the treatment of MDS prior to enrollment
* Performance status: Karnofsky ≥ 60%
* Adequate organ function defined as:
* Cardiac: LVEF at rest ≥ 35% (RIC cohort) or LVEF at rest ≥ 40% (FIC cohort), or LVFS ≥ 25%
* Pulmonary: DLCO, FEV1, FVC ≥ 50% predicted by pulmonary function tests (PFTs). DLCO value may be corrected or uncorrected for hemoglobin
* Hepatic: total bilirubin ≤ 2.5 mg/dL, and ALT, AST, and ALP < 5 x ULN (unless ALT, AST, and/or ALP are disease related)
* Renal: SCr within normal range for age (see table 5.1B). If SCr is outside normal range for age, CrCl > 40 mL/min/1.73m2 must be obtained (measured by 24-hour (hr) urine specimen or nuclear glomerular filtration rate (GFR), or calculated GFR (by Cockcroft-Gault formula)
* Subjects must have the ability to give informed consent according to applicable regulatory and local institutional requirements
* Availability of deceased HLA MMUD cryopreserved product through Ossium cryobank
* HLA MMUD defined as 4-7/8 HLA-allele matching at MHC class (A, B, or C) or MHC class II (DRB1)
* Additional MHC class II HLA (DP and DQ) typing will be collected, but not incorporated in donor selection

Exclusion Criteria:

* Pediatric patients (17 years or younger)
* Suitable HLA-matched related or 8/8 allele matched (HLA-A, -B, -C, -DRB1) unrelated donor excluding Ossium product
* Autologous HCT < 3 months prior to the time of signing the informed consent form
* Pregnancy or lactation
* Treatment with an investigational drug or other interventional GVHD clinical trials
* Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings)
* Prior allogeneic HCT
* Primary myelofibrosis or myelofibrosis secondary to essential thrombocythemia or polycythemia vera
* Subjects with MDS may not receive RIC and must be < 50 years of age at the time of signing the informed consent form
* Any condition(s) or diagnosis, both physical or psychological, or physical exam finding that in the investigator's opinion precludes participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Neutrophil engraftment | Day 35 Post HCT
  Run-in safety phase primary endpoint; Neutrophil engraftment is defined as neutrophil recovery by Day 35. Neutrophil recovery is defined as donor-derived absolute neutrophil count (ANC) ≥ 500/mm3 for three consecutive days with evidence of donor chimerism in bone marrow or peripheral blood. Full donor chimerism is >95%, and mixed donor chimerism is defined as 5-95%.
Cumulative incidence and kinetics of neutrophil and platelet recovery | Day 35 Post HCT
  Main phase primary endpoint; Neutrophil recovery is defined as achieving an absolute neutrophil count (ANC) greater than or equal to 500/mm3 for three consecutive measurements on three different days. The first of the three days will be designated the day of neutrophil recovery. The competing event is death without neutrophil recovery. For subjects who never drop ANC below 500/mm3, the date of neutrophil recovery will be Day 1 post-transplant. Platelet recovery is defined by two different metrics: the first day of a sustained platelet count greater than or equal to 20,000/mm3 or greater than or equal to 50,000/mm3 with no platelet transfusions in the preceding seven days. The first day of sustained platelet count above these thresholds will be designated the day of platelet engraftment. For subjects who never drop their platelet count below 20,000/mm3, the date of platelet recovery will be Day 1 post HCT.
Overall survival (OS) | 1-year Post HCT
  Main phase primary endpoint; The primary endpoint for the study is OS at 1-year post-HCT. The event is death from any cause. The time to this event is the time from HCT to death, loss to follow-up, or end of study (whichever comes first). Subjects who are lost to follow-up prior to 1-year will be censored at the time of the last observation, and the OS probability will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Cumulative incidences of aGVHD and cGVHD | 1-year Post HCT
  aGVHD is defined as any skin, gastrointestinal or liver abnormalities fulfilling the criteria of grades II-IV or grades III-IV. cGVHD is defined per National Institutes of Health (NIH) Consensus Criteria and includes organ involvement and severity, and overall global composite score (mild/moderate/severe).
Transplant-related mortality (TRM) | Day 100 and 1-year Post HCT
  TRM is defined as death without evidence of disease progression or recurrence. TRM will be evaluated at Day 100, 180, and 1-year (Day 365).
NK, B- and T-cell immune reconstitution | Days 35, 100, 180, and 1-year Post HCT
  Quantitative assessments of peripheral blood CD3, CD4, CD8, CD19 positive lymphocytes will be done through flow cytometric analysis at Days 35, 100, 180, and 365 post-HCT. Qualitative assessments will be tabulated according to time from transplant.
Progression free survival (PFS) | 1-year Post HCT
  Progression free survival will be estimated at 1-year (Day 365) post-transplant. An event for this time to event outcome is defined as disease relapse or progression, or death by any cause.
Event free survival (EFS) | 1-year Post HCT
  EFS will be estimated at 12 months post-HCT. An event for this time to event outcome includes graft failure (PGF by Day 35 or secondary graft failure), relapse or progression of underlying disease, death, grade III-IV acute GVHD, or NIH-severe chronic GVHD.
GVHD relapse free survival (GRFS) | 1-year Post HCT
  GRFS will be estimated at 1-year (Day 365) post-transplant. An event for this time to event outcome is defined as relapse or progression of underling disease, graft failure, grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, or death by any cause.
Cumulative incidence of cytokine release syndrome (CRS) | Day 14 Post HCT
  Overall incidence of CRS of any grade and grade 3 or 4 CRS post-transplant will be reported on all patients. CRS will be defined and graded using the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading criteria.
Donor chimerism | Days 35, 56, 100, 180, and 1-year Post HCT
  Peripheral blood chimerism (% of donor chimerism) in whole blood (unsorted) will be described on Day 35, 56, 100, 180, and 1-year (Day 365). Donor cell engraftment will be assessed with donor/recipient chimerism studies at Day 100. Chimerism may be assessed in CD3 blood cell fraction. For the purpose of this protocol, mixed chimerism is defined as the presence of donor cells, as a proportion of total cells to be less than 95% but at least 5% in the bone marrow or peripheral blood. Full donor chimerism is defined as greater than or equal to 95% of donor cells. Mixed and full chimerism will be evidence of donor cell engraftment. Donor cells of less than 5% by Day 35 will be considered as graft rejection. The proportion of patients with each level of chimerism described above will be described as part of this outcome. For sorted blood cell fractions, CD3+ donor cell chimerism will be used to define the donor/recipient chimerism status.
Cumulative incidences of viral reactivations and infections | Days 100, 180, and 1-year Post HCT
  The incidence of Cytomegalovirus (CMV), Epstein-Barr virus (EBV), BK virus, Adenovirus (ADV), and Human herpesvirus (HHV-6) viral activations and infections at Days 100, 180 and 1-year (Day 365).
Cumulative incidence of primary disease relapse/progression | 1-year Post HCT
  Testing for recurrent malignancy in the blood, bone marrow or other sites will be used to assess relapse and progression post-HCT. For the purpose of this study, relapse is defined by either morphological, cytogenetic/molecular or radiological evidence of disease consistent with pre-HCT features, in line with institutional standards. The event for this endpoint is the time interval from HCT to relapse/recurrence of disease or to last follow-up through 1-year (Day 365) post-HCT. Death in remission is considered a competing risk.

OTHER OUTCOMES:
Length of stay in hospital | Day 100 Post HCT
  Cumulative days alive and out of the hospital in the first 100 days and in the first year post-transplant.
Incidence of clinically-significant infections | 1-year Post HCT
  A clinically significant infection is defined as an infection that requires therapeutic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Auletta, MD, Study Chair — Center for International Blood and Marrow Transplant Research

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnstone BH, Woods JR, Goebel WS, Gu D, Lin CH, Miller HM, Musall KG, Sherry AM, Bailey BJ, Sims E, Sinn AL, Pollok KE, Spellman S, Auletta JJ, Woods EJ. Characterization and Function of Cryopreserved Bone Marrow from Deceased Organ Donors: A Potential Viable Alternative Graft Source. Transplant Cell Ther. 2023 Feb;29(2):95.e1-95.e10. doi: 10.1016/j.jtct.2022.11.010. Epub 2022 Nov 17. PMID 36402456